CLINICAL TRIAL: NCT06928233
Title: Association of the TNFAIP3 Genomic Locus With Immune-mediated TTP
Brief Title: Association of TNFAIP3 With Immune-mediated TTP
Acronym: A20iTTP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Principal Investigator, Ilaria Mancini, PhD, Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: A20iTTP; 2022-0469 (Other Grant/Funding Number: Fondazione Cariplo)
Record Dates: First submitted 2025-04-07; First posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Thrombotic Thrombocytopenic Purpura, Acquired
Keywords: A20; iTTP; TNFAIP3
MeSH Terms: conditions — Thrombotic thrombocytopenic purpura, acquired | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients with iTTP (Other): Intervention: blood sampling during standard collection for routine testing, with additional sample for experimental analyses.
  Interventions: Procedure: blood sampling
- Healthy donors (Other): Intervention: blood sampling during standard donation, with an additional sample collected for experimental analyses.
  Interventions: Procedure: blood sampling

INTERVENTIONS:
Procedure: blood sampling — Blood sampling for experimental analyses.

SUMMARY:
This study aims to investigate whether genetic variation in the TNFAIP3 locus is associated with immune-mediated thrombotic thrombocytopenic purpura (iTTP), and whether such association is mediated by decreased expression of A20 (TNFAIP3). The study includes a case-control design to assess genotype-expression association and a cohort study to evaluate clinical outcomes such as disease relapse.

ELIGIBILITY:
Patients:

Inclusion Criteria:

* Diagnosis of iTTP
* Above 12 years of age
* Caucasian, Italian origin
* Written informed consent to participate in the study

Exclusion Criteria:

* Patients who do not meet the above-listed criteria will be excluded from participation in the study.

Controls will be healthy Italian volunteers of Caucasian ethnicity, with no history of thrombotic thrombocytopenic purpura, frequency-matched to cases by age and sex, and who have provided written informed consent to participate in the study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-04-04 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Allele frequency of TNFAIP3 variants in cases vs controls | Baseline

SECONDARY OUTCOMES:
TNFAIP3 (A20) mRNA expression levels in peripheral blood | Baseline
  TNFAIP3 (A20) mRNA expression levels in peripheral blood of cases versus controls
Association between TNFAIP3 genotype and gene expression | Baseline
Clinical relapse rate of iTTP during follow-up | Baseline
  Association between TNFAIP3/A20 variation and iTTP relapse in iTTP patients
Severity of acute iTTP episodes | Baseline
  Association between TNFAIP3/A20 variation and the severity of acute iTTP (composite endpoint including death, treatment refractoriness, exacerbation, and prolonged disease course)
Age at iTTP onset | Baseline
  Association between TNFAIP3/A20 variation and age at onset in iTTP patients

CONTACTS AND LOCATIONS:
Overall Officials: Ilaria Mancini, PhD, Principal Investigator — Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Locations (1):
- Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico, Milan, Italy

IPD SHARING:
Plan to Share IPD: No